CLINICAL TRIAL: NCT06480305
Title: Effect Of Post Dinner Snack and Pre-Breakfast Consumption on Sleep Quality, Heart Rate Variability, Temperature, Interleukin-6, And Cortisol Levels in Healthy Males.
Brief Title: Impact of Evening Snacks and Pre-Breakfast Intake on Sleep, Heart Rate Variability, and Stress Markers in Healthy Males.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRC/24/1037 Humaira Fayyaz
Record Dates: First submitted 2024-06-05; First posted 2024-06-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Circadian Rhythm
Keywords: sleep; Heart Rate Variability; stress; cortisol; Interleukin-6; post dinner snack; prebreakfast; nuts

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Pre-breakfast and post dinner snack (A1) (Active Comparator): The Group A1 participants will not receive anything except for consuming a post-dinner snack. This is the control group for Prebreakfast and post-dinner snack groups.
  Interventions: Dietary Supplement: Post dinner snack
- Pre-breakfast and post dinner snack (A2) (Experimental): The Group A2 participants will consume post-dinner snacks consisting of 7-8 peanuts, one walnut, 2 cashews, 2 almonds, and 2 pistachios, and a prepackaged dose of 25 peanuts as a pre-breakfast snack.
  Interventions: Dietary Supplement: Post dinner snack; Dietary Supplement: Pre-Breakfast-1
- Pre-breakfast and post dinner snack (A3) (Experimental): The Group A3 participants will consume post-dinner snacks consisting of 7-8 peanuts, one walnut, 2 cashews, 2 almonds, and 2 pistachios, and a prepackaged dose of 25 raisins as a pre-breakfast snack.
  Interventions: Dietary Supplement: Post dinner snack; Dietary Supplement: Pre-Breakfast-2
- Pre-breakfast and post dinner snack (A4) (Experimental): The Group A4 participants will consume post-dinner snacks consisting of 7-8 peanuts, one walnut, 2 cashews, 2 almonds, and 2 pistachios, and a prepackaged dose of 5 peanuts on one day and 25 raisins as a pre-breakfast snack on the other day.
  Interventions: Dietary Supplement: Post dinner snack; Dietary Supplement: Pre-Breakfast-3
- Pre-breakfast but No Post dinner snack (B1) (No Intervention): The Group B1 participants will not receive anything not even pre-breakfast. This is the control group for Pre-breakfast and no post-dinner snacks.
- Pre-breakfast but No Post dinner snack (B2) (Experimental): The Group B2 participants will consume a prepackaged dose of 25 peanuts. Along with Pre-breakfast but no post-dinner snack.
  Interventions: Dietary Supplement: Pre-Breakfast-1
- Pre-breakfast but No Post dinner snack (B3) (Experimental): The Group B3 participants will consume a prepackaged dose of 25 raisins. Along with Pre-breakfast but No Post dinner snack.
  Interventions: Dietary Supplement: Pre-Breakfast-2
- Pre-breakfast but No Post dinner snack (B4) (Experimental): The Group A4 participants of the group will prepackaged dose of 25 peanuts one and the other day will consume 25 raisins. They alternate peanuts and raisins for the period of intervention. Along with Pre-breakfast but No Post dinner snack.
  Interventions: Dietary Supplement: Pre-Breakfast-3

INTERVENTIONS:
Dietary Supplement: Post dinner snack — one walnut, 2 cashews, 2 almonds, and 2 pistachios.
  Arms: Pre-breakfast and post dinner snack (A1); Pre-breakfast and post dinner snack (A2); Pre-breakfast and post dinner snack (A3); Pre-breakfast and post dinner snack (A4)
Dietary Supplement: Pre-Breakfast-1 — Prepackaged dose of 25 peanuts.
  Arms: Pre-breakfast and post dinner snack (A2); Pre-breakfast but No Post dinner snack (B2)
Dietary Supplement: Pre-Breakfast-2 — Prepackaged dose of 25 raisins
  Arms: Pre-breakfast and post dinner snack (A3); Pre-breakfast but No Post dinner snack (B3)
Dietary Supplement: Pre-Breakfast-3 — Prepackaged dose of 25 peanuts on one day and 25 raisins as a pre-breakfast.
  Arms: Pre-breakfast and post dinner snack (A4); Pre-breakfast but No Post dinner snack (B4)

SUMMARY:
The body has a natural 24-hour rhythm. This rhythm affects factors like body temperature, sleep and Heart Rate Variability (HRV). Dietary choices influence these physiological processes of the body. Poor sleep quality can increase stress and raise levels of a hormone called cortisol, affecting our heart and insulin levels. Heart rate variability (HRV) which is the time between heartbeats, is also influenced by sleep and the body's rhythm. Lower HRV levels have been linked to heart and mental health issues. Little research is present on the effects of post-dinner snacks and pre-breakfast interventions on sleep quality, Heart Rate Variability (HRV), temperature, Interleukin-6, and cortisol levels. It is hypothesised that eating a post-dinner snack and first pre-breakfast will affect sleep quality, heart rate variability, IL -6, cortisol levels and temperature in healthy males.

DETAILED DESCRIPTION:
The body's internal clock, circadian rhythms, works on a 24-hour cycle and is managed by a part of the brain called the hypothalamus. These rhythms control various bodily functions like temperature, hunger, emotions, and even our sleep-wake cycle. During sleep, hormones like cortisol, growth hormone, and insulin influence processes such as glucose metabolism. For instance, insulin levels drop while we sleep to allow the body to use stored energy, but rise again before waking. Poor sleep quality, even with adequate duration, can lead to increased stress and elevated cortisol levels, potentially affecting insulin and heart health. Heart rate variability (HRV), is the variation in time between heartbeats and is influenced by factors like stress, diet, and sleep quality. Lower HRV levels are associated with cardiovascular and mental health issues. Disruptions in the circadian sleep cycle can also affect the gut-brain axis, which involves communication between the gut and the brain via the vagus nerve. This axis influences gastrointestinal function and can impact inflammatory markers like interleukin-6 (IL-6), which in turn affect HRV and cardiovascular health. Dietary choices play a significant role in shaping the body's physiological processes. Nuts can positively impact HRV and sleep quality due to their nutrient content. A post-dinner snack consumed about three hours after dinner and a balanced pre-breakfast meal is important for maintaining stable blood sugar levels and overall health. Nuts, such as peanuts, almonds, cashews, pistachios, and walnuts, along with raisins, offer numerous health benefits. These contain fibre, protein, healthy fats, and essential nutrients that promote satiety, metabolic well-being, and digestive health. Thus this research aims to investigate the effects of post-dinner snacks and pre-breakfast interventions on HRV, sleep quality, IL-6, cortisol, and temperature. By exploring the relationship between dietary choices and physiological processes, we hope to gain insight into how to optimize health and well-being.

The participation will go through 2 assessments; at baseline and after intervention. For comparison two-way ANOVA followed by Post hoc-Tuckey test and for correlation between HRV and other parameters will be done using Pearson Correlation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No comorbidities like CVS, neurological, respiratory, liver and kidney diseases
* No skin allergy

Exclusion Criteria:

* Individuals with any comorbidities (Heart, liver , kidney, respiratory diseases)
* Individuals on any Medication
* Individuals with diagnosed insomnia
* Obese individual with BMI greater then 30
* Smokers
* Diagnosed patients with stress and anxiety
* Individuals with fever

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male adult participants will be taken to avoid the effect of hormone of female monthly cycle on HRV data
Enrollment: 80 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | Baseline
  The data will be collected from the Fitbit wristband and will be analyzed through the HRV time-domain, frequency domain methods.
  The values of high-frequency (HF) measure (power in the range of 0.15-0.4 Hz) will be considered normal. The values near 0.15Hz will be considered as reflecting sympathetic dominance and values of 0.4Hz will be considered good reflecting parasympathetic dominance. The low-frequency (LF) (power in the range: 0.04-0.15 Hz).
  VLF's Very Low-Frequency power band is between 0.003 Hz and 0.05 Hz. The LF/HF ratio reflects the balance between PNS and the sympathetic nervous system activity. The normal values are 2.2 ± 3.4
  Time domain measurements include:
  SDNN: values below 50 ms will be classified as unhealthy, values of 50-100 ms have compromised health, and above 100 ms are healthy RMSSD;RMSSD (ms) 20-89ms NN50:103.40 ms is the normal value. The values below 103.40 will be considered as high risk.
Heart Rate Variability | 3 weeks
  The data will be collected from the Fitbit wristband and will be analyzed through the HRV time-domain, frequency domain methods.
  The values of high-frequency (HF) measure (power in the range of 0.15-0.4 Hz) will be considered normal. The values near 0.15Hz will be considered as reflecting sympathetic dominance and values of 0.4Hz will be considered good reflecting parasympathetic dominance. The low-frequency (LF) (power in the range: 0.04-0.15 Hz).
  VLF's Very Low-Frequency power band is between 0.003 Hz and 0.05 Hz. The LF/HF ratio reflects the balance between PNS and the sympathetic nervous system activity. The normal values are 2.2 ± 3.4
  Time domain measurements include:
  SDNN: values below 50 ms will be classified as unhealthy, values of 50-100 ms have compromised health, and above 100 ms are healthy RMSSD;RMSSD (ms) 20-89ms NN50:103.40 ms is the normal value. The values below 103.40 will be considered as high risk.
Determination of sleep quality | Baseline
  For sleep, the Pittsburgh Sleep Quality Index (PSQI) a self-rated questionnaire, will be used to assess sleep quality.
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The sub-scores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Determination of sleep quality | 3 weeks
  For sleep, the Pittsburgh Sleep Quality Index (PSQI) a self-rated questionnaire, will be used to assess sleep quality.
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The sub-scores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Serum Cortisol | Baseline
  Quantitative determination of cortisol concentrations in serum will be done by using a cortisol ELISA Kit. The measurement will be done in the morning. range of serum cortisol in the morning is from 10 to 20 micrograms per deciliter. A serum level of 10 micrograms per deciliter will be considered as low levels and a serum level coming up to 20 micrograms per deciliter will be considered as high; the higher the level the higher the stress level.
Serum Cortisol | 3 weeks
  Quantitative determination of cortisol concentrations in serum will be done by using a cortisol ELISA Kit. The measurement will be done in the morning. range of serum cortisol in the morning is from 10 to 20 micrograms per deciliter. A serum level of 10 micrograms per deciliter will be considered as low levels and a serum level coming up to 20 micrograms per deciliter will be considered as high; the higher the level the higher the stress level.
Serum Interleukin-6 | Baseline
  Quantitative determination of interleukin-6 concentrations in serum will be done by using an interleukin-6 ELISA Kit. The measurement will be done in the morning. The level of Serum Interleukin-6 is from 7-18pg/ml. A serum level of 7 pg/ml of Serum Interleukin-6 will be considered low levels and a serum level coming to 18/ml will be considered as high; the higher the level the higher the stress level.
Serum Interleukin-6 | 3 weeks
  Quantitative determination of interleukin-6 concentrations in serum will be done by using an interleukin-6 ELISA Kit. The measurement will be done in the morning. The level of Serum Interleukin-6 is from 7-18pg/ml. A serum level of 7 pg/ml of Serum Interleukin-6 will be considered low levels and a serum level coming to 18/ml will be considered as high; the higher the level the higher the stress level.
Body Temperature | Baseline
  Participants will be instructed to record their body temperature before getting up from bed in the morning by a digital thermometer. the body temperature is considered normal between 97 F (36.1 C) and 99 F (37.2 C).
Body Temperature | 3 weeks
  Participants will be instructed to record their body temperature before getting up from bed in the morning by a digital thermometer. the body temperature is considered normal between 97 F (36.1 C) and 99 F (37.2 C).

SECONDARY OUTCOMES:
Blood pressure | Baseline
  Data will be collected from the Fitbit wristband. A blood pressure of 120/80 will be considered normal. A blood pressure of 130/ 85 will be considered high.
Blood pressure | 3 weeks
  Data will be collected from the Fitbit wristband. A blood pressure of 120/80 will be considered normal. A blood pressure of 130/ 85 will be considered high.
Heart rate | Baseline
  Data will be collected from Fitbit wrist band.
Heart rate | 3 weeks
  Data will be collected from Fitbit wrist band.
lipid profile | Baseline
  Data will be collected from blood samples. The optimal or target level for each part of the standard lipid test is listed below:
  Total cholesterol: Below 200 mg/dL HDL cholesterol: Above 60 mg/dL LDL cholesterol: Below 100 mg/dL Triglycerides: Below 150 mg/dL values of the Total cholesterol at 190-200 mg/dl will be considered as borderline and those greater than 210 will be considered as high.
  Values of HDL cholesterol Above 60 mg/dLwill be considered good and values lower than 60 mg/dL will be considered bad Values of LDL cholesterol lower than 100 mg/dL will be considered good and higher Values of more than 100 mg/dL will be considered as bad.
  Values of Triglycerides below 150 mg/dL will be considered good and higher than 150 mg/dL will be considered bad
lipid profile | 3 weeks
  Data will be collected from blood samples. The optimal or target level for each part of the standard lipid test is listed below:
  Total cholesterol: Below 200 mg/dL HDL cholesterol: Above 60 mg/dL LDL cholesterol: Below 100 mg/dL Triglycerides: Below 150 mg/dL values of the Total cholesterol at 190-200 mg/dl will be considered as borderline and those greater than 210 will be considered as high.
  Values of HDL cholesterol Above 60 mg/dLwill be considered good and values lower than 60 mg/dL will be considered bad Values of LDL cholesterol lower than 100 mg/dL will be considered good and higher Values of more than 100 mg/dL will be considered as bad.
  Values of Triglycerides below 150 mg/dL will be considered good and higher than 150 mg/dL will be considered bad
Short Multidimensional Inventory Lifestyle-SMILE C | baseline
  Multidimensional measure of lifestyle. It comprises 27 items. Answers are measured through a 4-point Likert scale, and scores are calculated by summing the responses (some questions have inverted score). The higher the SMILE score, the healthier the lifestyle pattern.
Short Multidimensional Inventory Lifestyle-SMILE C | 3 weeks
  Multidimensional measure of lifestyle. It comprises 27 items. Answers are measured through a 4-point Likert scale, and scores are calculated by summing the responses (some questions have inverted score). The higher the SMILE score, the healthier the lifestyle pattern.
Liver Function Test | baseline
  Data will be collected from blood samples. The optimal or target level for each part of the standard Liver test is listed below:
  Alanine aminotransferase(ALT): 7-55U/L Aspartate aminotransferase(AST):8-48U/L Alkaline phosphatase(ALP): 45-115U/L Bilirubin: less than1mg/dL Albumin3.4-5.4g/dL
  Values of Alanine aminotransferase(ALT) of 7 will U/L be considered normal and values of 55U/L will be considered high Aspartate aminotransferase(AST) value of8 U/L will be considered normal and 48U/L will be considered high Alkaline phosphatase(ALP) value of 45-U/L will be considered normal and 115 U/L will be considered high Bilirubin values of less than1mg/dL will be considered normal and more will be considered high Albumin values of 3.4 g/dL will be considered normal and more than 5.4 will be considered high
Liver Function Test | 3 weeks
  Data will be collected from blood samples. The optimal or target level for each part of the standard Liver test is listed below:
  Alanine aminotransferase(ALT): 7-55U/L Aspartate aminotransferase(AST):8-48U/L Alkaline phosphatase(ALP): 45-115U/L Bilirubin: less than1mg/dL Albumin3.4-5.4g/dL Values of Alanine aminotransferase(ALT) of 7 will U/L be considered normal and values of 55U/L will be considered high Aspartate aminotransferase(AST) value of8 U/L will be considered normal and 48U/L will be considered high Alkaline phosphatase(ALP) value of 45-U/L will be considered normal and 115 U/L will be considered high Bilirubin values of less than1mg/dL will be considered normal and more will be considered high Albumin values of 3.4 g/dL will be considered normal and more than 5.4 will be considered high
Renal function test | base line
  Data will be collected from blood samples. The optimal or target level for each part of the renal function tests are listed below:
  serum Urea: 2.5-6-5mmol/litre. Values of 2.5-mmol/litre will be considered normal and values of 6.5mmol/L and above will be considered high Serum creatinine: 0.7-1.4mmol/dL in males. Values of 0.7mmol/dLwill be considere normal and values of 1.4mmol/dL and above will be considered high
  Uric acid: 4-7 mmol/dL in males. Values of 4 mmol/litre will be considere normal. Values of 7 mmol/L and above will be considered high.
  Sodium : values of 135-145mmol/L will be considere normal. Values of 145mmol/L and above will be considered high Potassium: 3.5-5.0 mmol/dL values. These values will be considere normal and values of 5.0 mmol/dL and above will be considered high Calcium: 2.2-2.6 mmol/L. These will be considered normal and values of 2.7 mmol/L and above will be considered high Phosphate : 0.9-1.3 mmol/dlitre Chloride : 96-106 mmol/dL
Renal function test | 3 weeks
  Data will be collected from blood samples. The optimal or target level for each part of the renal function tests are listed below:
  serum Urea: 2.5-6-5mmol/litre. Values of 2.5-mmol/litre will be considered normal and values of 6.5mmol/L and above will be considered high Serum creatinine: 0.7-1.4mmol/dL in males. Values of 0.7mmol/dLwill be considere normal and values of 1.4mmol/dL and above will be considered high
  Uric acid: 4-7 mmol/dL in males. Values of 4 mmol/litre will be considere normal. Values of 7 mmol/L and above will be considered high.
  Sodium : values of 135-145mmol/L will be considere normal. Values of 145mmol/L and above will be considered high Potassium: 3.5-5.0 mmol/dL values. These values will be considere normal and values of 5.0 mmol/dL and above will be considered high Calcium: 2.2-2.6 mmol/L. These will be considered normal and values of 2.7 mmol/L and above will be considered high Phosphate : 0.9-1.3 mmol/dlitre Chloride : 96-106 mmol/dL
C reactive protein | base line
  will be done through the blood samples. The values are 0.3 to 1.0 mg/dL avalue of 0.3 will be considere normal and value of 1.0mg/dl and more will be considered elevated.
C reactive protein | 3 weeks
  will be done through the blood samples. The values are 0.3 to 1.0 mg/dL avalue of 0.3 will be considere normal and value of 1.0mg/dl and more will be considered elevated.
Depression Anxiety Stress Scales | base line
  It is a 21-item self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress. The DASS yields three subscale scores for depression, anxiety, and tension/stress. The lower the score the lower the symptoms the higher the score the higher the severity.
Depression Anxiety Stress Scales | 3 weeks
  It is a 21-item self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress. The DASS yields three subscale scores for depression, anxiety, and tension/stress. The lower the score the lower the symptoms the higher the score the higher the severity.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, Study Director — Riphah University
Locations (1):
- Imran Amjad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No